CLINICAL TRIAL: NCT01556776
Title: CLLM1-Protocol of the German CLL-Study Group (GCLLSG) A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of the Efficacy and Safety of Lenalidomide (Revlimid®) as Maintenance Therapy for High-risk Patients With Chronic Lymphocytic Leukemia Following First-line Therapy
Brief Title: A Study of Lenalidomide Maintenance for High-risk Patients With CLL Following First-line Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLLM1; 2011-004698-98 (EudraCT Number); RV-CLL-GCLLSG-0725 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2022-01-05 (Actual); Status verified 2021-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL; High Risk; Maintenance
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Experimental): lenalidomide maintenance following firstline treatment with FCR, BR, FR, or FC(if Rituximab is contraindicated)
  Interventions: Drug: lenalidomide
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lenalidomide — placebo or lenalidomide 5 mg daily on days 1-28 of the first 28-day cycle. If the 5 mg dose level is well tolerated, escalation to 10 mg daily on days 1-28 of cycle 2-6 is permitted; further escalations starting with the 7th cycle and up to the 12th cycle to 15 mg daily is permitted. If after 12 cycles of treatment subjects still present with MRD levels of ≥ 10-4 in peripheral blood and previous dose levels are well tolerated, starting with the 13th cycle up to progression 20 mg daily is permitted. If after 18 cycles of treatment for subjects still present with MRD.levels of ≥ 10-4 in peripheral blood and previous dose levels are well tolerated, starting with the 19th cycle up to progression 25 mg daily is permitted. 25 mg is the maximal daily dose of lenalidomide
  Other Names: Revlimid
  Arms: Lenalidomide
Drug: Placebo — placebo or lenalidomide 5 mg daily on days 1-28 of the first 28-day cycle. If the 5 mg dose level is well tolerated, escalation to 10 mg daily on days 1-28 of cycle 2-6 is permitted; further escalations starting with the 7th cycle and up to the 12th cycle to 15 mg daily is permitted. If after 12 cycles of treatment subjects still present with MRD levels of ≥ 10-4 in peripheral blood and previous dose levels are well tolerated, starting with the 13th cycle up to progression 20 mg daily is permitted. If after 18 cycles of treatment for subjects still present with MRD.levels of ≥ 10-4 in peripheral blood and previous dose levels are well tolerated, starting with the 19th cycle up to progression 25 mg daily is permitted. 25 mg is the maximal daily dose of lenalidomide
  Arms: Placebo

SUMMARY:
CLLM1 is a phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel-group study that compares the efficacy and safety of oral lenalidomide maintenance therapy to that of placebo maintenance therapy in high-risk subjects with Chronic Lymphocytic Leukemia (CLL) who have achieved at least a partial response (PR) and either:

* MRD levels of ≥ 10-2 or
* MRD levels of ≥ 10-4 - < 10-2 combined with at least one of the following factors:

  * an unmutated IGHV-status
  * 17p-deletion or
  * TP53 mutation after first line therapy with FCR, FR, BR or FC (in case of of contraindications to receive Rituximab).

DETAILED DESCRIPTION:
CLLM1 is a phase 3 multicenter, randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy and safety of lenalidomide administered as maintenance treatment to subjects with CLL who have responded to first-line therapy (induction) achieving a response of at least PR and are at high risk of early progression. This study will compare the efficacy of lenalidomide maintenance treatment versus placebo at prolonging progression free survival (PFS); and as secondary endpoints assess overall survival, the safety of lenalidomide treatment and evaluate Minimal residual disease (MRD) kinetics in peripheral blood whilst subjects are on maintenance.

Although maintenance therapy has been established in recent years for the treatment of a subset of subjects with Non-Hodgkin's Lymphoma (NHL), it is a novel concept in the management of CLL. It is not regularly used and only a limited number of small studies have been conducted evaluating consolidation/maintenance therapy for limited periods of time with alemtuzumab or rituximab. Based on the limited amount of available data, it appears that maintenance therapy may improve the quality of remission in CLL subjects and prolong progression-free survival (PFS). A large phase 3 trial investigating lenalidomide as maintenance following response to second line therapy is ongoing. However, a large well-controlled study has not been conducted to investigate the beneficial effect of maintenance therapy following front line therapy; specifically in subjects with aggressive disease. This phase 3 study will evaluate whether lenalidomide maintenance therapy will prolong PFS in CLL subjects with a high risk of early progression following first line treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must understand and voluntarily sign an informed consent form.
2. Age ≥ 18 years at the time of signing the informed consent form.
3. Must be able to adhere to the study visit schedule and other protocol requirements.
4. Must have a documented diagnosis of CLL (IWCLL guidelines for the diagnosis and treatment of chronic lymphocytic leukemia1.
5. Must have been treated with one of the first line induction therapies: fludarabine/cyclophosphamide, fludarabine/rituximab, fludarabine/cyclophosphamide/rituximab, pentostatin/cyclophosphamide/rituximab or bendamustine/rituximab.
6. Must have achieved a response of at least PR ((IWCLL guidelines for the diagnosis and treatment of chronic lymphocytic leukemia )following completion (minimum 4 cycles) of first line induction therapy prior to randomization, and have either:

   * MRD levels in the peripheral blood at final restaging of ≥10-2 or
   * MRD levels in the peripheral blood at final restaging of ≥10-4 - <10-2 combined with an unmutated IGHV-status or 17p-deletion or TP53 mutation.
7. Must have completed last cycle of at least 4 cycles of first-line induction no less than 8 weeks (56 days) and no greater than 20 weeks (140 days) prior to randomization.
8. Subjects who completed first-line induction treatment with less than 6 cycles but at least 4 cycles should document reason for early discontinuation.
9. Must have an Eastern Cooperative Oncology Group (ECOG see appendix 11.13) performance status score of ≤2.
10. Negative serological Hepatitis B test or negative PCR in case of positive serological test without evidence of an active infection, negative testing of Hepatitis C RNA, negative HIV test within 6 weeks prior to randomization.
11. Females of childbearing potential (FCBP)† must:

    * Have two negative medically supervised pregnancy tests prior to starting of study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices complete and continued sexual abstinence.
    * Either commit to continued abstinence from heterosexual intercourse (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, two reliable forms of effective contraception simultaneously to achieve a PEARL-Index <1 without without interruption (Highly effective methods: Intrauterine device (IUD), Hormonal (birth control pills, injections, implants), Tubal ligation, Partner's vasectomy, Additional effective methods: Male condom, Diaphragm, Cervical Cap). 28 days prior to starting study drug, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
12. Male subjects must:

    * Agree to use a condom during sexual contact with a FCBP, even if they have had a vasectomy, throughout study drug therapy, during any dose interruption and after cessation of study therapy.
    * Agree to not donate semen during study drug therapy and for a period after end of study drug therapy.
13. All subjects must:

    * Have an understanding that the study drug could have a potential teratogenic risk.
    * Agree to abstain from donating blood while taking study drug therapy and following discontinuation of study drug therapy.
    * Agree not to share study medication with another person.
    * Be counseled about pregnancy precautions and risks of fetal exposure.
14. Willingness to inform the general practitioner

Exclusion Criteria:

1. A CIRS Score of more than 6 or a single score of 4 for an organ system limiting the ability to receive an intensive treatment
2. Active infections requiring systemic antibiotics.
3. Systemic infection CTC grade 3 or 4 that has not resolved > 2 months prior to randomization in spite of adequate anti-infective therapy.
4. Autologous or allogeneic bone marrow transplant as first line therapy.
5. Pregnant or lactating females.
6. Systemic treatment for CLL in the interval between completing the last cycle of first-line induction therapy and randomization.
7. Participation in any clinical study or having taken any investigational therapy which would interfere with the study drug for a disease other than CLL within 28 days prior to initiating maintenance therapy.
8. Known presence of alcohol and/or drug abuse.
9. Central nervous system (CNS) involvement as documented by spinal fluid cytology or imaging. Subjects who have signs or symptoms suggestive of leukemic meningitis or a history of leukemic meningitis must have a lumbar puncture procedure performed within two weeks prior to randomization.
10. Prior history of malignancies, other than CLL, unless the subject has been free of the disease for ≥5 years. Exceptions include the following:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histological finding of prostate cancer (TNM stage of T1a or T1b)
11. History of renal failure requiring dialysis.
12. Prior therapy with lenalidomide.
13. Any of the following laboratory abnormalities:

    * Calculated (method of Cockcroft-Gault) creatinine clearance of <60 mL/min
    * Absolute neutrophil count (ANC) < 1,000/μL (1.0 X 109/L)
    * Platelet count < 50,000/μL (50 X 109/L)
    * Serum aspartate aminotransferase (AST)/serum glutamic-oxaloacetic transaminase (SGOT) or alanine transaminase (ALT)/serum glutamate pyruvate transaminase (SGPT) > 3.0 x upper limit of normal (ULN)
    * Serum total bilirubin > 2.0 mg/dL (with the exception of Gilbert's Syndrome)
14. Uncontrolled hyperthyroidism or hypothyroidism.
15. Venous thromboembolism within one year.
16. ≥ Grade-2 neuropathy.
17. Uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
18. Disease transformation (active) (i.e. Richter's Syndrome, prolymphocytic leukemia).
19. Known allergy to allopurinol if the subject has bulky disease.
20. Prisoners, or subjects who are institutionalized by regulatory or court order or persons who are who are in dependence to the sponsor or an investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) based on independent review committee | up to 6 years
  Time from the date of randomization to the date of first documented disease progression (as defined by the iWCLL response criteria, see section 4.11.1.2) or death by any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival (PFS) based on investigator's assessment | up to 6 years
  Time from the date of randomization to the date of first documented disease progression (as defined by the iWCLL response criteria, see section 4.11.1.2) or death by any cause, whichever occurs first.
Overall survival (OS) | up to 6 years
  Time from the date of randomization to the date of death due to any cause
Safety - adverse events (AEs) | up to 6 years
  Type, frequency and severity of adverse events (AEs) and relationship of AEs to lenalidomide or placebo; premature withdrawals
Miminimal residual disease (MRD) levels in peripheral blood (PB) | up to 6 years
  MRD levels assessed by quantitative highly sensitive flow cytometry (MRD flow) of the PB

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fink, MD, Study Chair — German CLL Study Group; Barbara Eichhorst, MD, Principal Investigator — German CLL Study Group
Locations (2):
- Germany (2):
  - University Hospital Cologne, Cologne
  - German CLL Study Group, Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fink AM, Bahlo J, Robrecht S, Al-Sawaf O, Aldaoud A, Hebart H, Jentsch-Ullrich K, Dorfel S, Fischer K, Wendtner CM, Nosslinger T, Ghia P, Bosch F, Kater AP, Dohner H, Kneba M, Kreuzer KA, Tausch E, Stilgenbauer S, Ritgen M, Bottcher S, Eichhorst B, Hallek M. Lenalidomide maintenance after first-line therapy for high-risk chronic lymphocytic leukaemia (CLLM1): final results from a randomised, double-blind, phase 3 study. Lancet Haematol. 2017 Oct;4(10):e475-e486. doi: 10.1016/S2352-3026(17)30171-0. Epub 2017 Sep 12. PMID 28916311
- [Result] Furstenau M, Fink AM, Schilhabel A, Weiss J, Robrecht S, Eckert R, de la Serna J, Crespo M, Coscia M, Vitale C, Bottcher S, Weppner G, Ritgen M, Stilgenbauer S, Tausch E, Fischer K, Hallek M, Eichhorst B, Bruggemann M, Herling CD. B-cell acute lymphoblastic leukemia in patients with chronic lymphocytic leukemia treated with lenalidomide. Blood. 2021 Apr 22;137(16):2267-2271. doi: 10.1182/blood.2020008609. No abstract available. PMID 33512465